CLINICAL TRIAL: NCT01007786
Title: The Ventricular Catheter Placement Study: Assessment of Efficacy and Safety of an Ultrasound Guided Shunt Insertion Technique
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 32371; HCRN 002 (Other: HCRN Protocol Number); 1RC1NS068943-01 (NIH)
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Pediatric Hydrocephalus
Keywords: Pediatric Hydrocephalus; Ultrasound Guided Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Shunt failure remains a significant problem in pediatric patients with hydrocephalus. If reliable techniques for the accurate placement of ventricular catheters can be developed, shunt survival may improve. The purpose of this study is to assess the efficacy and safety of the ultrasound guided shunt insertion technique in the hands of experienced surgeons. The primary outcome measure is ventricular catheter location determined from post-operative brain images. The study is being conducted by the Hydrocephalus Clinical Research Network (HCRN), a network established to conduct multi-institutional clinical trials on pediatric hydrocephalus. Pediatric neurosurgeons at HCRN centers enrolled in this study will perform either ultrasound guided shunt surgery or a conventional shunt surgery. Patients who undergo conventional shunt surgery will serve as a contemporary control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinical and radiographic evidence of hydrocephalus as determined by a pediatric neurosurgeon and require a ventriculoperitoneal shunt (atrial, pleural, gallbladder and other shunt systems are excluded)
* Patients can have no prior history of shunt insertion for hydrocephalus. A history of an external ventricular drain, subgaleal reservoir-catheter, or subgaleal shunt is permissible
* Patients must be less than 18 years of age at the time of shunt insertion

Exclusion Criteria:

* Active CSF or abdominal infection
* Spread of tumor in the subarachnoid space documented on enhanced imaging (CT or MRI) of the head or spine
* CSF leak without hydrocephalus
* Pseudotumor cerebri
* Dandy-Walker malformation or arachnoid cyst as a cause of hydrocephalus
* Loculations within the ventricular system
* Hydranencephaly, alobar holoprosencephaly or any other congenital anomaly of the brain that severely distorts the ventricular anatomy such that ventricular catheter location cannot be determined
* Other systemic disorders that would preclude the insertion/revision of a ventricular shunt
* Other difficulties that would preclude follow-up at one year (e.g. terminal illness with life expectancy less than 1 year)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric hydrocephalus patients undergoing first time shunt placement for hydrocephalus.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for the study is ventricular catheter location (VCL) as assessed on the first post-operative scan (US, CT, or MRI brain). | The first post-operative scan will only be used in the study if it occurs within 105 days of shunt insertion.

SECONDARY OUTCOMES:
Shunt survival will be reported. | Up to one year after the date of shunt placement.
Any complications, intraoperative and postoperative, will be reported. | From the time of surgery until the time the subject is discharged from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: William Whitehead, MD, MPH, Study Chair — HCRN, Texas Children's Hospital; Jay Riva-Cambrin, MD, Principal Investigator — HCRN, Primary Children's Medical Center; Abhaya Kulkarni, MD, PhD, Principal Investigator — HCRN, Sick Children's Hospital, Toronto, Ontario; Jay Wellons, MD, Principal Investigator — HCRN, Children's Hosptial of Alabama; John Kestle, MD, Principal Investigator — Chair, Hydrocephalus Clinical Research Network
Locations (4):
- United States (3):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
- Sick Children's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Whitehead WE, Riva-Cambrin J, Wellons JC 3rd, Kulkarni AV, Holubkov R, Illner A, Oakes WJ, Luerssen TG, Walker ML, Drake JM, Kestle JR; Hydrocephalus Clinical Research Network. No significant improvement in the rate of accurate ventricular catheter location using ultrasound-guided CSF shunt insertion: a prospective, controlled study by the Hydrocephalus Clinical Research Network. J Neurosurg Pediatr. 2013 Dec;12(6):565-74. doi: 10.3171/2013.9.PEDS1346. Epub 2013 Oct 11. PMID 24116981
- See also: Hydrocephalus Clinical Research Network — http://www.hcrn.org